CLINICAL TRIAL: NCT01670266
Title: A Double-masked, Placebo-controlled, Dose-escalation Study and Double-masked, Two-sequence, Crossover Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of ONO-9054 in Patients With Ocular Hypertension or Mild Open-Angle Glaucoma
Brief Title: Single and Multiple Dose Escalation and Two-sequence Crossover Study of ONO-9054 in Patients With Ocular Hypertension or Mild Open-angle Glaucoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ono Pharma USA Inc (Industry)
Responsible Party: Sponsor
Organization: Ono Pharmaceutical Co. Ltd (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ONO-9054IOU002
Record Dates: First submitted 2012-08-15; First posted 2012-08-22 (Estimated); Last update posted 2013-06-03 (Estimated); Status verified 2013-05

CONDITIONS: Ocular Hypertension (OHT); Mild Open Angle-glaucoma (OAG)
Keywords: ONO-9054; ocular hypertension; OHT; Open angle-glaucoma; OAG; Glaucoma; Eye diseases
MeSH Terms: conditions — Ocular Hypertension; Glaucoma, Open-Angle; Glaucoma; Eye Diseases | interventions — propan-2-yl 4-(6-(4-(2,5-difluorophenoxy)-3-hydroxybut-1-en-1-yl)-7-hydroxyoctahydro-2H-cyclopenta(b)oxepin-3-yl)butanoate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Experimental Arm 1 (Experimental): Experimental Eye drops 3.0 µg/mL QD both eyes on Day 1, 5-18
  Interventions: Drug: ONO-9054
- Experimental Arm 2 (Experimental): Experimental Eye drops 10.0 µg/mL QD both eyes on Day 1, 5-18
  Interventions: Drug: ONO-9054
- Experimental Arm 3 (Experimental): Experimental Eye drop 30.0 µg/mL QD both eyes on day 1, 5-18
  Interventions: Drug: ONO-9054
- Experimental Arm 4 (Experimental): Experimental Eye drop, 2 sequence crossover Cohort [1 dose; 1-30 µg/mL]to be determined and placebo
  Interventions: Drug: ONO-9054; Drug: Placebo
- Placebo Arm (Placebo Comparator): Matched placebo eye drops dosed in same manner as ONO-9054
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ONO-9054
  Arms: Experimental Arm 1; Experimental Arm 2; Experimental Arm 3; Experimental Arm 4
Drug: Placebo
  Arms: Experimental Arm 4; Placebo Arm

SUMMARY:
The primary objective of this study is to evaluate the safety and tolerability of 3 planned doses of ONO-9054 in the eyes of adult male and female patients with ocular hypertension (OHT) or mild open angle-glaucoma (OAG).

The secondary objectives are to evaluate Pharmacodynamics (PD) and to characterize the pharmacokinetic (PK) profile of ONO-9054 and its metabolite in plasma and to compare its tolerability following morning and evening dosing.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects age 18-80 (inclusive) with confirmed diagnosis of OHT or OAG
* Confirmed diagnosis of bilateral OHT or chronic open-angle glaucoma
* Able to undergo washout of all ocular drugs
* An IOP ≥ 22mmHg at 8:00 AM and ≥ 21 mmHg at 10:00 AM in at least one eye; but ≤ 35 mmHg at all time points in both eyes on Day -2 and Day -1
* Central corneal thickness 500-600 µm at screening in both eyes
* BCVA 20/100 or better in both eyes

Exclusion Criteria:

* Any history of severe ocular trauma in either eye at any time
* Any history of previous intraocular or ocular laser surgery within the past 3 months or any refractive surgery procedure within the past 6 months of screening visit in the study eye(s)
* Cataracts that prevent observation of the fundus in either eye

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-08; Primary Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of ONO-9054 | up to 14 days
  Safety and tolerability of ONO-9054 will be measured using vital signs, ECGs, laboratory tests, ocular exams, physical examination and incidence/severity of adverse events over a dosing period of up to 14 days

SECONDARY OUTCOMES:
Characterization of PK profiles | up to 14 days
  The mean concentrations of ONO-9054 and its active metabolite will be measured in plasma in order to determine peak and trough levels over a dosing period of 14 days
Evaluation of PD measurements | up to 14 days
  The pharmacodynamic measurement will be intraocular pressure. Relative changes with respect to baseline will be assessed after 14 days of administration under both AM and PM dosing conditions.
Comparison of safety, tolerability between once daily morning and once daily evening | 14 days
  Safety and tolerability of a single concentration will be evaluated by review of adverse events and any change from baseline in ocular symptoms in a crossover arm in which the active drug is administered for 14 days under both AM and PM dosing conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Ono Pharma USA, Inc., Study Director — Ono Pharmaceutical Co. Ltd
Locations (3):
- United States (3):
  - Costa Mesa Clinical Site, Costa Mesa, California
  - Newport Beach (satellite site), Newport Beach, California
  - Santa Ana (satellite site), Santa Ana, California

REFERENCES:
- [Derived] Berlin MS, Rowe-Rendleman C, Ahmed I, Ross DT, Fujii A, Ouchi T, Quach C, Wood A, Ward CL. EP3/FP dual receptor agonist ONO-9054 administered morning or evening to patients with open-angle glaucoma or ocular hypertension: results of a randomised crossover study. Br J Ophthalmol. 2016 Jun;100(6):843-7. doi: 10.1136/bjophthalmol-2015-307000. Epub 2015 Oct 9. PMID 26453641